CLINICAL TRIAL: NCT01174810
Title: An Open Label, Single Site, 12 Month, Phase II, Randomised Controlled Trial Evaluating the Safety and Efficacy of Exendin-4 (Exenatide) in the Treatment of Patients With Moderate Severity Parkinson's Disease.
Brief Title: Exendin-4 as a Treatment for Parkinson's Disease - Pilot Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University College, London (Other)
Responsible Party: Dr Thomas Foltynie, UCL
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09/0391; 2009-018137-37 (EudraCT Number)
Record Dates: First submitted 2010-08-02; First posted 2010-08-04 (Estimated); Last update posted 2012-03-23 (Estimated); Status verified 2012-03

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; PD; Moderate Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Exenatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention)
- Exenatide (Experimental)
  Interventions: Drug: Exenatide

INTERVENTIONS:
Drug: Exenatide — Exenatide, 5 micrograms twice a day for 1 month and 10 micrograms twice a day for 11 months. Total duration of treatment 12 months
  Other Names: Byetta; Exendin-4
  Arms: Exenatide

SUMMARY:
Exenatide is a licensed, safe and effective treatment for patients with Diabetes mellitus. Laboratory work has shown strong, reproducible evidence that this drug has beneficial "disease modifying" effects when given to animals with a range of experimental models of Parkinson's disease (PD). This project aims to make an initial evaluation of possible benefits of Exenatide among patients with moderate symptoms of PD. The drug will be given as a twice daily 10microgram injection under the skin in a similar way to one of the conventional "symptomatic" treatments for PD (Apomorphine).

Forty patients with moderate symptoms of PD will be recruited and randomised to receive Exenatide injections twice daily, or to act as controls in this open label trial. Detailed assessments will be made of all patients at baseline and periodically for a total of 14 months. The primary outcome measure will be the change between baseline and follow up, in the severity of a validated PD assessment scale (the UPDRS part 3 motor score) after an overnight period free of conventional PD medication. Secondary measures will include adverse event reports, self completed questionnaires, and blood test results. Aside from these assessments, all patients will continue their regular PD medications throughout the trial with adjustments made only according to clinical need.

In a subgroup of patients (n=10), brain scans that assess the severity of PD, will be performed at both baseline and follow up to help understand possible mechanisms of action of Exenatide.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Idiopathic Parkinson's disease of moderate severity- equivalent to Hoehn/ Yahr stage 2 to 2.5 (Bilateral symptoms but still physically independent).

Male or female. Female patients to be post menopausal (defined as 12 months of spontaneous amenorrhoea or 6 months spontaneous amenorrhoea with FSH levels greater than 40mIU/ml), surgically sterilised (post hysterectomy and/or oophorectomy). Male patients with female partners that have child bearing potential must use adequate contraception (condoms +/-spermicidal gel/foam) throughout the duration of the trial period.

* Age 45-70 years
* Disease onset after age 40 years
* Disease duration > 5 years
* On L-dopa treatment. Patient must be on oral L-dopa treatment - with or without dopamine agonist including Apomorphine, MAO-B inhibitor, COMT inhibitor, Amantadine, Beta blocker, anticholinergic treatment History of wearing off phenomena- duration of action of single dose of L-dopa < 6 hours Stable PD medication for preceding 3 months- i.e. no change in medication type or dose.
* UPDRS motor off medication score >15
* L-dopa responsiveness. Defined as >33% improvement in UPDRS motor off medication score following L-dopa challenge
* Able to give informed consent
* Able to comply with trial protocol and willing to attend necessary clinic visits off medication.

Exclusion Criteria:

* Diagnosis or suspicion of other cause for parkinsonism including Vascular parkinsonism, post traumatic parkinsonism, drug or toxin induced parkinsonism, or other neurodegenerative condition including Multiple System Atrophy, Progressive Supranuclear Palsy, Huntington's disease, Wilson's disease, Pantothenate kinase Neurodegeneration (PKAN), Alzheimer's disease, Creutzfeld Jacob disease.
* Known abnormality on CT or MRI brain imaging considered to be causing symptoms or signs of neurological dysfunction, or considered likely to compromise compliance with trial protocol.

Concurrent dementia defined by a score lower than 120 on the Mattis Dementia Rating Scale.

* Concurrent severe depression defined by a score greater than 16 on the MADRS Exposure to neuroleptic drugs within 6 months prior to baseline assessment Prior intracerebral surgical intervention for Parkinson's disease including Deep Brain stimulation, lesional surgery, growth factor administration, gene therapy or cell transplant
* Already actively participating in a trial of a device, drug or surgical treatment for Parkinson's disease, or trial participation within previous 30 days.
* Type 1 Diabetes mellitus
* Type 2 Diabetes mellitus on insulin treatment
* End stage renal disease or severely impaired renal function with creatinine clearance <30ml/min
* History of severe cardiac disease (Angina, Myocardial infarction or cardiac surgery in preceding 2 years)
* History of pancreatitis
* History of alcoholism
* Severe gastrointestinal disease including gastroparesis
* Ongoing treatment with sulphonylurea
* Females that are pregnant or breast feeding or of child bearing potential.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-07; Primary Completion 2013-03 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to 12 months & 14 months between patients on active Exenatide treatment and PD controls in respect of their UPDRS-off-medication motor subscore.

SECONDARY OUTCOMES:
Adverse event profile among patients treated with Exenatide compared with matched PD controls. Change from baseline to 12 months/ 14 months between patients on active treatment and PD controls in respect of list given below
  * the UPDRS on medication motor subscore
  * the UPDRS ADL subscore
  * dyskinesia rating scale
  * timed motor tests
  * the Mattis Dementia rating scale
  * the Montgomery & Asberg Depression rating scale
  * the PDQ39
  * the EQ-5D
  * the NMS Quest
  * the SCOPA Sleep scale
  * the SCOPA AUT scale
  * the Smell Identification test
  * DAT (SPECT) scan appearances.

CONTACTS AND LOCATIONS:
Locations (1):
- National Hospital for Neurology and Neurosurgery, London, United Kingdom

REFERENCES:
- [Derived] Aviles-Olmos I, Dickson J, Kefalopoulou Z, Djamshidian A, Ell P, Soderlund T, Whitton P, Wyse R, Isaacs T, Lees A, Limousin P, Foltynie T. Exenatide and the treatment of patients with Parkinson's disease. J Clin Invest. 2013 Jun;123(6):2730-6. doi: 10.1172/JCI68295. PMID 23728174